CLINICAL TRIAL: NCT04841681
Title: Effectiveness of Video-based Psychotherapy in Reducing Distress in Patients With COVID-19 Treated in a Hospital Isolation Ward in Jakarta
Brief Title: Video-based Psychotherapy for COVID-19 Patients in Isolation Ward in Jakarta
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Collaborators: National Institute of Health Research and Development, Ministry of Health Republic of Indonesia (Other)
Responsible Party: Principal Investigator, Petrin Redayani Lukman, Principal Investigator, Indonesia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 20-05-0546
Record Dates: First submitted 2021-04-06; First posted 2021-04-12 (Actual); Last update posted 2021-04-12 (Actual); Status verified 2021-04

CONDITIONS: Covid19; Distress, Emotional
Keywords: COVID-19; distress; patients in isolation wards; video-based psychotherapy
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: This study utilized the quasi-experimental design with a pre-test-post-test and without a control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Video-based Psychotherapy (Experimental): The group received the intervention of video-based psychotherapy.
  Interventions: Behavioral: Video-based Psychotherapy

INTERVENTIONS:
Behavioral: Video-based Psychotherapy — Participants in the group watched three short videos. Therapeutic elements in the three consecutive short videos included relaxation therapy, managing thoughts and feelings, and mindfulness. Each video has a duration of just over 10 minutes.
  In the first video, the participants were introduced to the purpose and benefits of relaxation techniques. These included rhythmic breathing techniques, progressive muscle relaxation, imagining a comforting and quiet place, and positive self-talk. In the second video about managing thoughts and feelings, the participants were introduced to the notion of acceptance of their condition. They were invited to recognize the emergence of negative feelings and thoughts related to acceptance. In the last video about mindfulness, patients were introduced to three basic mindfulness skills: observation, elaboration, and participation.

SUMMARY:
The COVID-19 pandemic has made severe impact worldwide for those inflicted by the disease, the caretakers, the general public, as well as the health care system. Hospitalized patients with COVID-19 experience physical isolation during treatment. Isolation may lead to psychological distress that could negatively affect well-being such as affective states of depression, anxiety, and loneliness. Thus, creative ways to deliver psycho-social support are needed when face-to-face therapy sessions may not possible. We investigated the effectiveness of video-based psychotherapy in reducing distress in patients with COVID-19 treated in a general hospital isolation ward in Jakarta. This study included 42 patients with COVID-19, who were asked to watch three brief psychotherapy videos about relaxation, managing thoughts and emotions, and mindfulness. Before and after watching the videos, patients were asked to complete the Subjective Units of Distress Scale (SUDS) to measure their stress level. 31 subjects experienced a significant decrease in SUDS score after the intervention. Our brief video-based psychotherapy intervention may have a positive effect on reducing distress in hospitalized COVID-19 patients in areas with scarce resources.

DETAILED DESCRIPTION:
The coronavirus disease 2019 (COVID-19) pandemic has brought severe consequences worldwide. Indonesia is one of the countries which has been affected by this pandemic. The examination, treatment, and monitoring of individuals with COVID-19 often requires them to be in a hospital isolation ward. There are a lot of factors which could negatively affect the mental health of such patients during their isolation, to the point that they develop significantly debilitating conditions.

Several psychotherapy interventions have been known to be effective during a pandemic situation. The interventions include those based on techniques of relaxation, managing thoughts and feelings, and mindfulness. These methods could help reducing negative and catastrophic thoughts about the future, reducing distress level and hyperarousal, and other beneficial effect. However, due to the high transmission rate of SARS-CoV-2 virus (severe acute respiratory syndrome-coronavirus 2), face-to-face therapy sessions are rendered difficult to hold under the circumstances. Thus, we conducted a pilot study to test the impact of a video-based psychotherapy intervention on distress and well-being in hospitalized COVID-19 patients in a medical isolation ward.

This pilot study included 42 patients with COVID-19, aged 20-59. Participants watched three brief psychotherapy videos covering relaxation, managing thoughts and emotions, and mindfulness. Before and after watching the videos, patients were asked to complete the Subjective Units of Distress Scale (SUDS). 31 subjects experienced a significant median decrease in SUDS score after the intervention. The effect size was 0.485, with a 95% confidence interval of 0.302 to 0.634. Our brief video-based psychotherapy intervention may have a positive effect on reducing distress in hospitalized COVID-19 patients in areas with scarce resources. This study could be used as a reference for future studies regarding the method of choice for delivering psychotherapy intervention for patients in isolation ward during the COVID-19 pandemic.

ELIGIBILITY:
Inclusion Criteria:

* Patients with COVID-19 in Kiara Ultimate CMH (Cipto Mangunkusumo Hospital) isolation ward who are at least 18 years old
* Patients with COVID-19 in Kiara Ultimate CMH isolation ward who are able to give an informed consent
* Patients with COVID-19 in Kiara Ultimate CMH isolation ward who agreed to watch the psychotherapy videos about relaxation, managing thoughts and feelings, and mindfulness using electronic devices provided by the research team or their own devices independently

Exclusion Criteria:

* Patients in unstable conditions such as patients on a ventilator, experiencing breathing difficulties, or in need of oxygen support, with fluctuating levels of consciousness
* Patients with physical and intellectual disabilities that may hinder ability to understand instructions of the video-based psychotherapy intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2020-06-07 (Actual); Primary Completion 2020-08-25 (Actual); Study Completion 2020-08-26 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Subjective Units of Distress (SUDS) at Right After Receiving Video-based Psychotherapy | Baseline (before receiving the intervention of video-based psychotherapy) and immediately after receiving the intervention of video-based psychotherapy (right after the participants have finished watching the 30 minutes-long psychotherapy videos)
  Subjective Units of Distress (SUDS) is a self-rating instrument used to measure the distress level of an individual in a numeric scale from the scale of 0 (no distress) to 10 (extreme distress).
  Change = score right after participants have received the video-based psychotherapy - baseline score before they received the video-based psychotherapy

CONTACTS AND LOCATIONS:
Locations (1):
- dr. Cipto Mangunkusumo National General Hospital, Jakarta Pusat, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: Yes
We plan to share the data of participants' (identities will be initials only) demographic data and SUDS score before and after watching the video.
Time Frame: 1 month after publication.
Access Criteria: The data will be available through request to Petrin Redayani Lukman MD as the contact person, e-mail ptrn1010@yahoo.com.

REFERENCES:
- [Background] Abad C, Fearday A, Safdar N. Adverse effects of isolation in hospitalised patients: a systematic review. J Hosp Infect. 2010 Oct;76(2):97-102. doi: 10.1016/j.jhin.2010.04.027. PMID 20619929
- [Background] Zandifar A, Badrfam R, Yazdani S, Arzaghi SM, Rahimi F, Ghasemi S, Khamisabadi S, Mohammadian Khonsari N, Qorbani M. Prevalence and severity of depression, anxiety, stress and perceived stress in hospitalized patients with COVID-19. J Diabetes Metab Disord. 2020 Oct 29;19(2):1431-1438. doi: 10.1007/s40200-020-00667-1. eCollection 2020 Dec. PMID 33145259
- [Background] Brooks SK, Webster RK, Smith LE, Woodland L, Wessely S, Greenberg N, Rubin GJ. The psychological impact of quarantine and how to reduce it: rapid review of the evidence. Lancet. 2020 Mar 14;395(10227):912-920. doi: 10.1016/S0140-6736(20)30460-8. Epub 2020 Feb 26. PMID 32112714
- [Background] Zarghami A, Farjam M, Fakhraei B, Hashemzadeh K, Yazdanpanah MH. A Report of the Telepsychiatric Evaluation of SARS-CoV-2 Patients. Telemed J E Health. 2020 Dec;26(12):1461-1465. doi: 10.1089/tmj.2020.0125. Epub 2020 Jun 11. PMID 32525755
- [Background] Cheng W, Zhang F, Hua Y, Yang Z, Liu J. Development of a psychological first-aid model in inpatients with COVID-19 in Wuhan, China. Gen Psychiatr. 2020 Jun 17;33(3):e100292. doi: 10.1136/gpsych-2020-100292. eCollection 2020. PMID 32596642
- [Background] Sherifali D, Ali MU, Ploeg J, Markle-Reid M, Valaitis R, Bartholomew A, Fitzpatrick-Lewis D, McAiney C. Impact of Internet-Based Interventions on Caregiver Mental Health: Systematic Review and Meta-Analysis. J Med Internet Res. 2018 Jul 3;20(7):e10668. doi: 10.2196/10668. PMID 29970358
- [Background] Nelson NA, Bergeman CS. Daily Stress Processes in a Pandemic: The Effects of Worry, Age, and Affect. Gerontologist. 2021 Feb 23;61(2):196-204. doi: 10.1093/geront/gnaa187. PMID 33186445
- [Background] Nwachukwu I, Nkire N, Shalaby R, Hrabok M, Vuong W, Gusnowski A, Surood S, Urichuk L, Greenshaw AJ, Agyapong VIO. COVID-19 Pandemic: Age-Related Differences in Measures of Stress, Anxiety and Depression in Canada. Int J Environ Res Public Health. 2020 Sep 1;17(17):6366. doi: 10.3390/ijerph17176366. PMID 32882922
- [Result] Wei N, Huang BC, Lu SJ, Hu JB, Zhou XY, Hu CC, Chen JK, Huang JW, Li SG, Wang Z, Wang DD, Xu Y, Hu SH. Efficacy of internet-based integrated intervention on depression and anxiety symptoms in patients with COVID-19. J Zhejiang Univ Sci B. 2020 May;21(5):400-404. doi: 10.1631/jzus.B2010013. Epub 2020 Apr 1. PMID 32425006
- [Result] Liu K, Chen Y, Wu D, Lin R, Wang Z, Pan L. Effects of progressive muscle relaxation on anxiety and sleep quality in patients with COVID-19. Complement Ther Clin Pract. 2020 May;39:101132. doi: 10.1016/j.ctcp.2020.101132. Epub 2020 Mar 6. PMID 32379667
- [Result] Dekker RL, Moser DK, Peden AR, Lennie TA. Cognitive therapy improves three-month outcomes in hospitalized patients with heart failure. J Card Fail. 2012 Jan;18(1):10-20. doi: 10.1016/j.cardfail.2011.09.008. Epub 2011 Nov 9. PMID 22196836
- [Result] Conversano C, Di Giuseppe M, Miccoli M, Ciacchini R, Gemignani A, Orru G. Mindfulness, Age and Gender as Protective Factors Against Psychological Distress During COVID-19 Pandemic. Front Psychol. 2020 Sep 11;11:1900. doi: 10.3389/fpsyg.2020.01900. eCollection 2020. PMID 33013503
- [Result] Behan C. The benefits of meditation and mindfulness practices during times of crisis such as COVID-19. Ir J Psychol Med. 2020 Dec;37(4):256-258. doi: 10.1017/ipm.2020.38. Epub 2020 May 14. PMID 32406348
- [Result] Grazzi L, Rizzoli P, Andrasik F. Effectiveness of mindfulness by smartphone, for patients with chronic migraine and medication overuse during the Covid-19 emergency. Neurol Sci. 2020 Dec;41(Suppl 2):461-462. doi: 10.1007/s10072-020-04659-0. PMID 32794128
- [Result] Reyes AT. A Mindfulness Mobile App for Traumatized COVID-19 Healthcare Workers and Recovered Patients: A Response to "The Use of Digital Applications and COVID-19". Community Ment Health J. 2020 Oct;56(7):1204-1205. doi: 10.1007/s10597-020-00690-9. Epub 2020 Aug 9. No abstract available. PMID 32772205

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-20): https://cdn.clinicaltrials.gov/large-docs/81/NCT04841681/Prot_SAP_000.pdf